CLINICAL TRIAL: NCT06955533
Title: Single Dose Versus Double Dose Tamsulosin 0.4 and Solifenacin 5 in Management of Stent Related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hisham Arafa, H arafa, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MS23/ 2023
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-04

CONDITIONS: Stent Related Symptoms
MeSH Terms: interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double dose tamsulosin ans solifenacin (Active Comparator)
  Interventions: Drug: Double dose tamsulosin and solifenacin
- Single dose tamsulosin and solifenacin (Active Comparator)
  Interventions: Drug: Single dose tamsulosin and solifenacin

INTERVENTIONS:
Drug: Double dose tamsulosin and solifenacin — Odd number
  Arms: Double dose tamsulosin ans solifenacin
Drug: Single dose tamsulosin and solifenacin — Even number
  Arms: Single dose tamsulosin and solifenacin

SUMMARY:
This study was a randomized clinical trial conducted on 64 Egyptian patients from the outpatient clinic at Ain Shams University Hospital over a six-month period from 3/2024 to 9/2024.The study population was randomized into 2 groups. Group A included 32 patients with stent related symptoms receiving double doses of tamsulosin (Tamsulin® 0.4 mg 2 capsules taken together per day) and Solifenacin 10mg (Sofenacin® 10mg tab taken once daily).Group B included 32 patients with stent related symptoms receiving a standard dose of tamsulosin (0.4 mg once daily) and solifenacin (5 mg once daily).

ELIGIBILITY:
Inclusion Criteria:

- We included patients older than18 years of age, with presence of a double-J (DJ) stent in place, suffering from lower urinary tract symptoms (LUTS).Patients younger than 18 years of age, patients with a history of prostate or bladder surgery, lower urinary tract procedures, cancer, neurological conditions, pelvic radiation, diabetes, kidney dysfunction (acute or chronic), a solitary kidney, congenital urinary anomalies, or those taking medications such as α-blockers, beta-blockers, calcium channel blockers, 5-alpha reductase inhibitors, PDE5 inhibitors, anticholinergics, or nitrates were excluded. Additionally, patients with cardiac issues, residual stone fragments after surgery, multiple or bilateral ureteral stones, long-term or bilateral stents requiring frequent changes, interstitial cystitis, chronic cystitis, prostatitis, pregnant or breastfeeding women, and those unavailable for follow-up were also excluded from the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Improvement of ussq | 2 weeks
  This is a pilot study aiming to evaluate the effectiveness of Double dose versus standard dose of tamsulosin with solifenacin in relieving stent related symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt